CLINICAL TRIAL: NCT06911801
Title: In Vitro Study of [18F]F-FAPI-74 Feasibility in Vulvar Cancer
Acronym: FAPI_VULVA_1
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7284
Record Dates: First submitted 2025-02-12; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Vulvar Squamous Cell Carcinoma
Keywords: Vulvar Squamous Cell Carcinoma; FAPI; Phosphor imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Vulvar squamous cell carcinoma specimens obtained from surgical biopsies, stored in optimal cutting temperature compound and formalin-fixed paraffin-embedded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Tumour specimens stored both in optimal cutting temperature compound and formalin-fixed paraffin-embedded from patients with a first diagnosis of vulvar squamous cell carcinoma. Upon sectioning, the specimens will be analysed using phosphor imaging with FAPI radiopharmaceutical.

SUMMARY:
This study aims to investigate the expression of FAP by phosphor imaging in invasive vulvar squamous cell carcinoma specimens. This in vitro study will include all consecutive tumour specimens stored both in optimal cutting temperature (OCT) compound and formalin-fixed paraffin-embedded (FFPE) from patients with a first diagnosis of vulvar squamous cell carcinoma who underwent surgery at Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy.

DETAILED DESCRIPTION:
Vulvar cancer is a rare gynaecological tumour, affecting 2.5 out of 100,000 women per year. The most common histological type is squamous cell carcinomas. Current guidelines suggest 2-[18F]fluoro-2-deoxy-D-glucose ([18F]FDG) PET/CT for T2 or larger tumours or when metastases are suspected, even though few studies showed controversial results on small series about the diagnostic accuracy of [18F]FDG PET/CT for vulvar cancer. The recently developed fibroblast activation protein inhibitor (FAPI), labelled with gallium-68 or fluorine-18, may be a promising diagnostic tool for gynaecological cancers in the field of PET/CT imaging. There is an unmet need to characterize FAP expression at the whole-body level, to assess target expression for disease detection and FAP-directed therapies. This study aims to investigate the expression of FAP by phosphor imaging in vulvar squamous cell carcinoma specimens on OCT compound and FFPE sections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of invasive vulvar cancer with squamous cell histotype, both from primary tumour site and excised metastatic LNs.
* Availability of both FFPE and OCT stored samples from each primary tumour site and (when available) from the corresponding metastatic groin lymph nodes.
* Samples stored in sufficient quantity not to be completely exhausted by their use for this study.
* Optimal stored sample
* Available clinical and histopathological data

Exclusion Criteria:

- Coexistence of primary tumours other than vulvar cancer

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The specimens of patients with vulvar squamous cell carcinoma, who underwent surgery at the Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy, during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of specimens with FAP expression | 10 months
  Defines the proportion of VSCC specimens with expression of FAP (%).
Quantitative FAP binding | 10 months
  Quantitative FAP binding, measured as counts per minute (cpm)/mm2 of residual radioactivity after incubation time/washing step.
FAP binding affinity | 10 months
  FAP binding affinity, measured as % inhibition of specific binding plotted against the concentration of radiotracers.
Distribution of radiotracer in VSCC specimens | 10 months
  Distribution of radiotracer in VSCC specimens, measured as cpm/mm2 in specific regions of the specimens (e.g., hypoxic region, perivascular).

SECONDARY OUTCOMES:
Correlating FAP Expression in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Patients's Age | 10 months
  Probability of testing the correlation of FAP expression level (unit: digital light unit) with age (unit: years).
Correlating FAP Expression in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor FIGO Stage | 10 months
  Probability of testing the correlation of FAP expression level (unit: digital light unit) with tumor FIGO stage (adimensional).
Correlating FAP Expression in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor Pathological Grading | 10 months
  Probability of testing the correlation of FAP expression level (unit: digital light unit) with tumor pathological grading 1-2 vs 3 (adimensional).
Correlating FAP Expression in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor Pathological Histotype | 10 months
  Probability of testing the correlation of FAP expression level (unit: digital light unit) with tumor pathological histotype squamous vs other (adimensional).
Correlating FAP Expression in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor Morphology on Hematoxylin and Eosin Staining | 10 months
  Probability of testing the correlation of FAP expression level (unit: digital light unit) with tumor morphology on hematoxylin and eosin staining (H&E) (adimensional).
Correlating FAP Binding in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Patients's Age | 10 months
  Probability of testing the correlation of quantitative FAP binding (adimensional) with age (unit: years).
Correlating FAP Binding in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor FIGO Stage | 10 months
  Probability of testing the correlation of quantitative FAP binding (adimensional) with tumor FIGO stage (adimensional).
Correlating FAP Binding in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor Pathological Grading | 10 months
  Probability of testing the correlation of quantitative FAP binding (adimensional) with tumor pathological grading 1-2 vs 3 (adimensional).
Correlating FAP Binding in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor Pathological Histotype | 10 months
  Probability of testing the correlation of quantitative FAP binding (adimensional) with tumor pathological histotype squamous vs other (adimensional).
Correlating FAP Binding in Vulvar Squamous Cell Carcinoma Specimen (Derived by Phosphor Imaging With [18F]F-FAPI-74) to Tumor Morphology on Hematoxylin and Eosin Staining | 10 months
  Probability of testing the correlation of quantitative FAP binding (adimensional) with tumor morphology on hematoxylin and eosin staining (H&E) (adimensional).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Collarino, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klebermass EM, Dengler A, Weissenbock V, Ricken G, Wadsak W, Viernstein H, Hacker M, Mitterhauser M, Philippe C. Autoradiography on deparaffinized tissue sections - A feasibility study with 68Ga-labeled PET-tracers. Appl Radiat Isot. 2022 Nov;189:110425. doi: 10.1016/j.apradiso.2022.110425. Epub 2022 Aug 18. PMID 36030760
- [Background] Kalluri R. The biology and function of fibroblasts in cancer. Nat Rev Cancer. 2016 Aug 23;16(9):582-98. doi: 10.1038/nrc.2016.73. PMID 27550820
- [Background] Lindner T, Giesel FL, Kratochwil C, Serfling SE. Radioligands Targeting Fibroblast Activation Protein (FAP). Cancers (Basel). 2021 Nov 16;13(22):5744. doi: 10.3390/cancers13225744. PMID 34830898
- [Background] Oonk MHM, Planchamp F, Baldwin P, Mahner S, Mirza MR, Fischerova D, Creutzberg CL, Guillot E, Garganese G, Lax S, Redondo A, Sturdza A, Taylor A, Ulrikh E, Vandecaveye V, van der Zee A, Wolber L, Zach D, Zannoni GF, Zapardiel I. European Society of Gynaecological Oncology Guidelines for the Management of Patients with Vulvar Cancer - Update 2023. Int J Gynecol Cancer. 2023 Jul 3;33(7):1023-1043. doi: 10.1136/ijgc-2023-004486. PMID 37369376